CLINICAL TRIAL: NCT00854555
Title: The ATLET Study: Can Subjects With Incomplete Spinal Cord Injury Learn to Walk? A Randomized Clinical Trial
Brief Title: The ATLET Study: Can Subjects With Incomplete Spinal Cord Injury Learn to Walk?
Acronym: ATLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Norway Rehabilitation Center (Other)
Collaborators: Sunnaas Rehabilitation Hospital (Other); Norwegian School of Sport Sciences (Other); University of Tromso (Other); University of Oslo (Other); Norwegian Foundation for Health and Rehabilitation (Other); Norwegian Department of Health and Social Affairs (Other Government); Loma Linda University (Other)
Responsible Party: Principal Investigator, Synnove Knutsen, MD, PhD, Professor, North Norway Rehabilitation Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 980924076; P REK 69/2008; P REK 2009-634 (Other: National Committee for Medical and Health Research Ethics)
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury
Keywords: incomplete spinal cord injury; locomotor activity; walking function; gait
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- robot (Experimental): 30 persons with incomplete SCI who live within driving distance to Oslo and who meet the inclusion/exclusion criteria will be selected for randomization to robotic assisted training or control (conventional treatment). Intervention consists of locomotor training with robot for 60 days during 6 months period in an out-patient setting. Minimum 60 min training up to 3 times per week. Control group receives conventional training/treatment.
  Interventions: Other: Locomotor training with robot
- manual assistance (Experimental): 30 persons with incomplete SCI who live outside driving distance to Oslo and who meet inclusion/exclusion criteria will be selected for manually assisted training in Tromsø or control (conventional treatment). Intervention consists of 60 days locomotor training with manual assistance during 6 months period in an in-patient setting. Training 2 times per day total 120 minutes. Control group receives conventional training/treatment.
  Interventions: Other: Locomotor training with manual assistance

INTERVENTIONS:
Other: Locomotor training with robot — 60 days locomotor training during 6 months period in out-patient setting. Minimum 60 min training up to 3 times per week. Control group receives conventional training/treatment.
  Other Names: LOKOMAT
  Arms: robot
Other: Locomotor training with manual assistance — 60 days training during 6 months period on in-patient setting. Training 2 times per day total 120 minutes. Control group receives conventional training/treatment.
  Other Names: Vigor Equipment treadmill and suspension system; Therapist assisted
  Arms: manual assistance

SUMMARY:
The ATLET study will assess the effect of manual or robotic body-weight supported locomotor training of patients with stable motor incomplete spinal cord injury (SCI) on gait and overall ADL function as well as on estimated health care costs.

DETAILED DESCRIPTION:
There are approximately 100 new cases of spinal cord injuries (SCI) each year in Norway. Most of the SCI occur after traumatic accidents among young people and adults during the time of their productive life. Loss of walking and standing ability restricts their independent mobility and autonomy and severely impacts their quality of life.

The study has two arms: 1) manual locomotor training (Tromsø) and 2) robot assisted training (Oslo). Each study arm has 30 patients, randomized to receive standard care or intervention. The intervention group receives 60 days of intensive locomotor training over 6 months. Single-blind, before/after evaluation of effect will be performed at Sunnaas hospital using a standardized set of evaluation tools.

ELIGIBILITY:
Inclusion Criteria:

* Motor incomplete SCI grade AIS-C or -D
* Age: 18 - 70 years
* Body mass index of <30
* Wheelchair dependent
* At least 2 years since time of injury
* Cognitively unaffected and motivated for locomotor training
* Lives within driving distance of Oslo (< 70 km), if considered for the outpatient arm of the study.

Exclusion Criteria:

* Complete SCI grade AIS-A or -B
* Cognitively reduced
* BMI ≥ 30
* Age: under 18 years or above 71 years
* Spasms and contractures which can prevent locomotor training
* Changes in use of spasm reducing medication during intervention
* Significant osteoporosis in spine and/or joints
* Pregnancy (adequate contraceptive use is required of women in fertile age)
* Physical limitations for the use of the robotic orthosis
* Participation in other intensive training programs
* Those who live 70 or more kilometers from the Oslo training center, will be enrolled in the Tromso arm of the study.
* Other medical condition which can interfere with the training protocol
* Previous knee- or hip replacement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
To assess whether locomotor training with body-weight support in patients with motor incomplete SCI results in full or partial recovery of the ability to walk and/or stand. | 2-4 weeks before and after intervention
Patients with motor incomplete SCI are able to improve ADL function after locomotor training. | 2 - 4 weeks before and after intervention
Locomotor training is cost-effective rehabilitation. | 2-4 weeks before and after intervention

SECONDARY OUTCOMES:
Locomotor training in persons with motor incomplete SCI will lead to change in walking function | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in ADL function and independency | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in balance | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in strength in lower extremities | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in sensibility below the level of injury | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in ASIA impairment scale | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in quality of life | 2-4 weeks before and after intervention
Locomotor training in persons with motor incomplete SCI will lead to change in use of personal assistant or home health nurse | 2-4 weeks before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Synnove F Knutsen, MD PhD, Principal Investigator — North Norway Rehabilitation Center; Raymond Knutsen, MD MPH, Study Chair — ATLET Steering group; Nils Hjeltnes, MD PhD, Principal Investigator — Sunnaas Hospital
Locations (2):
- Norway (2):
  - Sunnaas Hospital, Oslo
  - North Norway Rehabilitation Center, Tromsø

REFERENCES:
- [Derived] Piira A, Lannem AM, Gjesdal K, Knutsen R, Jorgensen L, Glott T, Hjeltnes N, Knutsen SF, Sorensen M. Quality of life and psychological outcomes of body-weight supported locomotor training in spinal cord injured persons with long-standing incomplete lesions. Spinal Cord. 2020 May;58(5):560-569. doi: 10.1038/s41393-019-0401-2. Epub 2019 Dec 17. PMID 31848443